CLINICAL TRIAL: NCT01680809
Title: Compliance of Compression Therapy in Healed Venous Ulcerations
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CWCT-001
Record Dates: First submitted 2012-08-31; First posted 2012-09-07 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Venous Insufficiency
Keywords: Venous insufficiency; Venous stasis ulcerations; Compression stockings; Compression stocking compliance
MeSH Terms: conditions — Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Compression stocking 15-20mmHg (Experimental): Compression stocking 15-20mmHg
  Interventions: Device: Compression stocking 15-20mmHg
- Compression stocking 20-30mmHg (Experimental): Compression stocking 20-30mmHg
  Interventions: Device: Compression stocking 20-30mmHg

INTERVENTIONS:
Device: Compression stocking 15-20mmHg — Compression stocking with 15-20mmHg of compression
  Arms: Compression stocking 15-20mmHg
Device: Compression stocking 20-30mmHg — Compression stocking with 20-30mmHg of compression
  Arms: Compression stocking 20-30mmHg

SUMMARY:
This study seeks to determine if compliance with compression therapy is increased in patients with healed venous insufficiency ulcerations when lower levels of compression therapy are prescribed. This study will measure compliance with compression therapy at low levels of compression. It will also seek to determine if compression therapy aids in the prevention of venous insufficiency ulcer recurrence.

DETAILED DESCRIPTION:
This study looks to determine if patients with a history of venous insufficiency and recently healed venous insufficiency ulcerations are compliant with lower levels of compression therapy. It also seeks to evaluate the efficacy of compression therapy in the prevention of recurrence of venous insufficiency ulcerations.

ELIGIBILITY:
Inclusion Criteria:

* Recently healed venous insufficiency ulcerations
* History of venous insufficiency
* Patient from UH Richmond Wound Care Center (recently discharged/healed venous ulcerations)

Exclusion Criteria:

* Children
* Patients with diagnosed arterial insufficiency or ABI less than 0.5
* Patients that are diagnosed with Congestive Heart Failure and not cardiac cleared
* Patients with paralysis or incapacitated physically or mentally (due to inability to apply compression stockings)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Compliance of Compression Therapy | 12 months
  Patients will be assessed for compliance of compression therapy at the following intervals (1 month, 3 months, 6 months, 9 months, and 12 months) -- this will be accomplished via patient questionnaire/interview at scheduled appointments at each stated interval.

SECONDARY OUTCOMES:
Ulceration recurrence | 12 months
  We will evaluate if venous ulcerations have recurred with compression therapy over the course of 12 months. The patient will be seen/evaluated at appointments scheduled at 1 month, 3 months, 6 months, 9 months and 12 months. At each visit, the patient will be evaluated for recurrence of ulcerations. If ulceration recurs, then the patient will be removed from the study and be eligible for treatment of ulcerations.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole E Allen-Wilson, DPM, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- Richmond Medical Center (University Hospitals of Cleveland), Richmond Heights, Ohio, United States

REFERENCES:
- [Background] Milic DJ, Zivic SS, Bogdanovic DC, Karanovic ND, Golubovic ZV. Risk factors related to the failure of venous leg ulcers to heal with compression treatment. J Vasc Surg. 2009 May;49(5):1242-7. doi: 10.1016/j.jvs.2008.11.069. Epub 2009 Feb 23. PMID 19233601
- [Background] Gillespie DL; Writing Group III of the Pacific Vascular Symposium 6; Kistner B, Glass C, Bailey B, Chopra A, Ennis B, Marston B, Masuda E, Moneta G, Nelzen O, Raffetto J, Raju S, Vedantham S, Wright D, Falanga V. Venous ulcer diagnosis, treatment, and prevention of recurrences. J Vasc Surg. 2010 Nov;52(5 Suppl):8S-14S. doi: 10.1016/j.jvs.2010.05.068. Epub 2010 Aug 3. No abstract available. PMID 20678885
- [Background] Marston WA, Carlin RE, Passman MA, Farber MA, Keagy BA. Healing rates and cost efficacy of outpatient compression treatment for leg ulcers associated with venous insufficiency. J Vasc Surg. 1999 Sep;30(3):491-8. doi: 10.1016/s0741-5214(99)70076-5. PMID 10477642
- [Background] Nelson EA, Harper DR, Prescott RJ, Gibson B, Brown D, Ruckley CV. Prevention of recurrence of venous ulceration: randomized controlled trial of class 2 and class 3 elastic compression. J Vasc Surg. 2006 Oct;44(4):803-8. doi: 10.1016/j.jvs.2006.05.051. PMID 17012004
- [Background] Barwell JR, Davies CE, Deacon J, Harvey K, Minor J, Sassano A, Taylor M, Usher J, Wakely C, Earnshaw JJ, Heather BP, Mitchell DC, Whyman MR, Poskitt KR. Comparison of surgery and compression with compression alone in chronic venous ulceration (ESCHAR study): randomised controlled trial. Lancet. 2004 Jun 5;363(9424):1854-9. doi: 10.1016/S0140-6736(04)16353-8. PMID 15183623
- [Background] Baranoski S, Ayello EA. Wound Care Essentials: Practice Principles, 3rd ed. Philadelphia, PA: Lippincott Williams and Wilkins, 2011. Print.